CLINICAL TRIAL: NCT06219317
Title: Immunotherapy Consolidation After Radical Treatment of Synchronous Oligo-metastatic NSCLC
Acronym: ICARS
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: European Organisation for Research and Treatment of Cancer - EORTC (Network)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: EORTC-2029-LCG
Record Dates: First submitted 2024-01-03; First posted 2024-01-23 (Actual); Last update posted 2025-07-16 (Actual); Status verified 2025-07

CONDITIONS: NSCLC Stage IV
Keywords: NSCLC; cemiplimab; immunotherapy; oligometastatic disease; radical treatment
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung | interventions — cemiplimab

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Cemiplimab (Experimental): Cemiplimab IV 350 mg every 3 weeks for up to 12 months or until progression or discontinuation
  Interventions: Drug: Cemiplimab
- Placebo (Placebo Comparator): Placebo (saline solution) IV every 3 weeks for up to 12 months or until progression or discontinuation
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Cemiplimab — Cemiplimab is provided in a 10 ml glass vial
  Arms: Cemiplimab
Drug: Placebo — standard saline solution
  Arms: Placebo

SUMMARY:
This is a multi-center, double-blind, placebo-controlled randomized phase II study to assess whether continuation of cemiplimab treatment (for up to 12 months) increases progression-free survival (PFS) as compared to placebo in patients with a stage IV, synchronous, oligometastatic non-small cell lung cancer (NSCLC) who have not progressed following 4 cycles of cemiplimab with our without platinum-based chemotherapy and radical treatment.

Eligible patients are randomized with a 1:1 ratio to either the cemiplimab or placebo group and will undergo disease assessment (e.g. imaging, blood tests) at regular follow-up visits.

ELIGIBILITY:
1. Registration phase

   Inclusion criteria
   * Histologic or cytologic confirmation of NSCLC. If small-cell elements present, participant will be ineligible.
   * Synchronous oligometastatic disease at diagnosis - and still oligometastatic at registration into the study - defined as maximum 5 metastases, in maximum 3 organs. Hilar, mediastinal and/or supraclavicular lymph nodes are not considered as metastases.
   * Age at registration ≥18 years
   * Eastern Cooperative Oncology Group performance status (ECOG PS)/ World Health Organization (WHO) 0-1.
   * Hepatic function:
   * Serum total bilirubin ≤1.5x upper limit of normal (ULN), or ≤3x ULN, if liver metastases or in patients with history of Gilbert syndrome
   * Aspartate aminotransferase (AST) and/or alanine aminotransferase (ALT) ≤3x ULN (or ≤5x ULN, if liver metastases)
   * Renal function:
   * Glomerular filtration rate (GFR) based on the modification of diet in renal disease (MDRD) equation ≥30 mL/min
   * Bone marrow function:
   * Hemoglobin ≥9.0 g/dL
   * Absolute neutrophil count (ANC) ≥1.5 x 109/L
   * Platelet count ≥100 x 109/L
   * Women of childbearing potential (WOCBP) must have a negative serum or highly sensitive urine pregnancy test within 7 days prior to the first dose of treatment.

   Note: Women of childbearing potential are defined as premenopausal females capable of becoming pregnant (i.e., females who have had any evidence of menses in the past 12 months, with the exception of those who had prior hysterectomy). However, women who have been amenorrhoeic for 12 or more months are still considered to be of childbearing potential if the amenorrhea is possibly due to prior chemotherapy, antiestrogens, low body weight, ovarian suppression, or other reasons.
   * Patients of childbearing / reproductive potential should agree to use adequate birth control measures, as defined by the protocol, during the study treatment period and for:
   * At least 6 months after the last dose of pemetrexed-if pemetrexed was administered.
   * At least 6 months after the last dose of cemiplimab/placebo. A highly effective method of birth control is defined as a method which results in a low failure rate (i.e., less than 1% per year) when used consistently and correctly. Such methods are detailed in Appendix Y.
   * Women who are breast feeding should discontinue nursing prior to the first dose of study treatment and until:
   * At least 6 months after the last dose of pemetrexed, if pemetrexed was administered.
   * At least 6 months after the last dose of cemiplimab/placebo.
   * Capable of giving signed informed consent which includes compliance with the requirements and restrictions listed in the informed consent form (ICF) and in this protocol.

   Exclusion criteria
   * Presence of malignant pleural, pericardial and/or peritoneal effusion.
   * Presence of leptomeningeal carcinomatosis.
   * Tumour known to be positive for EGFR exon 19 or 21 mutations, ALK translocations or ROS1 fusions.
   * Prior pneumonectomy, radiotherapy (including mediastinal radiotherapy), chemotherapy, immune-check inhibitors or targeted therapy for lung cancer within the last 3 years before registration.
   * Previously treated brain metastases that are radiologically non-stable.

   Notes:
   * Patients with previously treated brain metastases, i.e., without evidence of progression for at least 4 weeks by repeat imaging (note that the repeat imaging should be performed during study screening), clinically stable and without requirement of steroid treatment for at least 14 days prior to first dose of study intervention, can participate. These treated brain metastasis will count as metastasis in the definition of oligometastatic disease.
   * Symptomatic brain metastases should be treated with surgery and/or stereotactic radiotherapy/ radiosurgery as soon as possible after diagnosis. If surgery is considered it must be applied before enrolment. Radiotherapy can be performed at any time.
   * History of any solid or hematological malignancy in the past 3 years before registration.

   Exceptions include patients who underwent successful definitive treatment of basal or squamous cell carcinoma of the skin, or any in-situ carcinoma(s).
   * Any uncontrolled, intercurrent illness or clinical situation that would, in the judgment of investigator, limit compliance with study requirements.
   * Any uncontrolled active infection, defined as an infection ≥ grade 3 according to CTCAE version 5.0.
   * Any autoimmune disease that has required systemic treatment in the past 2 years (defined as any use of disease modifying agents, corticosteroids or immunosuppressive drugs).

   Replacement therapy (e.g., thyroxine for hypothyroidism or insulin for type I diabetes) is not considered a form of systemic treatment.

   The following treatments are allowed:
   * Intranasal, inhaled and topical steroids as well as local steroid injections (e.g., intra articular injection).
   * Systemic corticosteroids at physiologic doses not to exceed 10 mg/day of prednisone or its equivalent.
   * Systemic corticosteroid replacement therapy for adrenal or pituitary insufficiency.
   * Steroids as premedication for hypersensitivity reactions (e.g., CT scan premedication)

     * Known active hepatitis B or C, defined as a positive HBV surface antigen (HBsAg) result or positive HCV RNA.
     * Known active HIV infection, defined as >200 copies of HIV per ml of blood.
     * History of interstitial lung disease (e.g., idiopathic pulmonary fibrosis, organizing pneumonia) or history of non-infectious pneumonitis that required systemic glucocorticoids to assist with management.

   A history of radiation pneumonitis in the radiation field is permitted as long as pneumonitis resolved ≥12 months prior to registration.

   • Immunosuppressive corticosteroid doses (>10 mg prednisone daily or equivalent) within 2 weeks prior to the first dose of cemiplimab.

   Patients who require brief courses of steroids (e.g., as prophylaxis for imaging studies due to hypersensitivity to contrast agents) can be included.
   * Participation in any other clinical study involving an investigational drug or device within 4 weeks before registration.
   * History of documented allergic reaction or acute hypersensitivity reaction attributed to antibody treatments.
   * Sensitivity to any of the study interventions, or components thereof, or other allergy that, in the opinion of the investigator, contraindicates participation in the study.
   * Any psychological, familial, sociological or geographical condition potentially hampering compliance with the study protocol, understanding and completion of questionnaires and follow-up schedule; those conditions should be assessed and discussed with the patient before the enrolment in the trial
2. At randomization Prior to treatment allocation for the consolidation phase an additional set of selection criteria need to be met and stratification factors provided.

Inclusion criteria

* Stable disease, partial or complete response according to RECIST v.1.1 after 4 cycles of induction treatment and radical treatment of all residual disease (if applicable). Patients with progressive disease will be excluded.
* Anticipated life expectancy >12 weeks
* Hepatic function:
* Serum total bilirubin ≤1.5x ULN (or ≤3x ULN, if liver metastases or in patients with history of Gilbert syndrome)
* AST and/or ALT ≤3x ULN (or ≤5x ULN, if liver metastases)
* Renal function:
* GFR based on MDRD equation ≥30 mL/min
* Bone marrow function:
* Hemoglobin ≥9.0 g/dL
* ANC ≥1.5 x 109/L
* Platelet count ≥100 x 109/L
* WOCBP must have a negative serum or highly negative urine pregnancy test within 7 days prior to the first dose of consolidation treatment.

Exclusion criteria

• Use of immunosuppressive corticosteroid doses (>10 mg prednisone daily or equivalent) within 2 weeks prior to the first dose of cemiplimab/placebo. Patients who require brief courses of steroids (e.g., as prophylaxis for imaging studies due to hypersensitivity to contrast agents) can be included.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 136 (Estimated)
Dates: Start 2025-01-14 (Actual); Primary Completion 2030-01 (Estimated); Study Completion 2030-01 (Estimated)

PRIMARY OUTCOMES:
Progression-free survival (PFS) | 9 years from first patient randomized
  PFS is defined as the time from the date of randomization until first occurrence of any of the following events:
  * Disease progression at any site: loco-regional progression/recurrence (related to primary tumour); progression/recurrence of oligometastatic lesions initially present at registration
  * Development of new metastatic lesions
  * Death due to any cause.
  Disease progression will be assessed using the RECIST 1.1 criteria.

SECONDARY OUTCOMES:
Overall survival (OS) | 6 years from first patient randomized
  OS is defined as the time from the date of randomization until date of death, for any reason
Time to disease progression | 6 years from first patient randomized
  Time to disease progression is defined as the time from the date of randomization to the date of first occurrence of any of the following events:
  * Disease progression at any site: loco-regional progression/recurrence (related to primary tumour); progression/recurrence of oligometastatic lesions initially present at registration
  * Development of new metastatic lesions
  * Death due to progressive disease.
Time to development of new metastatic lesions | 6 years from first patient randomized
  Time to development of new metastatic lesions is the time interval from the date of randomization to the date of first occurrence of any of the following events:
  * Development of new metastatic lesions not initially present at registration,
  * Death due to progressive disease.
Time to progression in oligometastatic lesions initially present at registration | 6 years from first patient randomized
  Time to progression in oligometastatic lesions initially present at registration is the time interval from the date of randomization to the date of first progression/recurrence in at least one of the oligometastatic lesions initially present at registration
AEs according to NCI-CTCAE v5.0 and SAEs | 9 years from first patient randomized
  This study will use the International Common Terminology Criteria for Adverse Events (CTCAE), version 5.0, for adverse event reporting
Patient reported QoL as measured by the EORTC QLQ-C30 questionnaire | 9 weeks from last patient last treatment
  This questionnaire is composed of 30 individual questions that are scored into 15 multi-item and single-item scales according the EORTC scoring manual. These include five functional scales (physical, role, emotional, social, and cognitive), nine symptom scales (fatigue, nausea and vomiting, pain, dyspnoea, insomnia, appetite loss, constipation, diarrhoea and financial difficulties) and a global health status/QoL scale.
  The functional and symptom questions follow the same structure using a 4-point Likert scale with responses from "not at all" to "very much".
  The questions on global health an QoL use a 7-point Likert scale with responses from "very poor" to "excellent".
Patient reported QoL as measured by the IL316 questionnaire - self assessment of treatment side effects | 9 weeks from last patient last treatment
  This questionnaire includes self-assessment of treatment side effects, most notable pneumonitis.
  The questions follow the same structure using a 4-point Likert scale with responses from "not at all" to "very much" and are scored according to the scale structure of their respective source questionnaire.
Patient reported QoL as measured by the IL316 questionnaire - questions from EORTC QLQ-LC29 questionnaire | 9 weeks from last patient last treatment
  This questionnaire includes 8 questions from the EORTC lung cancer specific module (QLQ-LC29) were selected: the coughing domain scale (2 questions), the dyspnoea scale (3 questions), chest pain (1 question) and physical capabilities (1 question).
  The questions follow the same structure using a 4-point Likert scale with responses from "not at all" to "very much" and are scored according to the scale structure of their respective source questionnaire.
Patient reported QoL as measured by the IL316 questionnaire - questions from EORTC QLQ-ELD14 questionnaire | 9 weeks from last patient last treatment
  This questionnaire includes 1 item from the validated QLQ-ELD14 questionnaire to include self-assessment on treatment burden: "How much has your treatment been a burden to you?" The questions follow the same structure using a 4-point Likert scale with responses from "not at all" to "very much" and are scored according to the scale structure of their respective source questionnaire.

OTHER OUTCOMES:
Tumour molecular profile (NGS panel, WES (including germline), RNAseq) | 6 years from first patient randomized
  FFPE tumour tissue will be collected at diagnosis, at metastasectomy and at progression (if available).
  NGS panel, WES (including germline), RNAseq will be used for analysis.
ctDNA analysis | 6 years from first patient randomized
  Blood will be collected at registration, at induction (C2D1), after induction, after radical therapy, at consolidation (every 9 weeks from C1D1 (5 times), at end of treatment and at PD.
Circulating biomarkers such as cytokines, or auto-Ab | 6 years from first patient randomized
  Blood will be collected at registration, at induction (C2D1), after induction, after radical therapy, at consolidation (every 9 weeks from C1D1 (5 times), at end of treatment and at PD.
Biomarker assessment of the tumour microenvironment | 6 years from first patient randomized
  FFPE tumour tissue and blood will be collected on regular time points during the study.
  Analysis will be using multiplex Immuno-Fluorescence (mIF) or other imaging techniques, and/or spatial transcriptomics.

CONTACTS AND LOCATIONS:
Overall Officials: Dirk de Ruysscher, MD, Study Chair — Maastro Clinic - Maastricht Radiation Oncology, Maastricht, Netherlands; Frank Aboubakar Nana, MD, Study Chair — Cliniques Universitaires Saint-Luc, Brussels, Belgium
Locations (17):
- Belgium (3):
  - Cliniques Universitaires Saint-Luc, Brussels
  - CHU Helora Pole Hospitalier Jolimont, Haine-Saint-Paul
  - CHU Mont Godinne - UCL Namur, Yvoir
- France (3):
  - CH de La Cote Basque - Saint Leon, Bayonne
  - Institut Paoli-Calmettes, Marseille
  - Groupe Hospitalier Paris Saint Joseph, Paris
- Italy (6):
  - ASST Ovest Milanese - Legnano, Legnano
  - Azienda Unita Locale Socio-Sanitaria N. 9-Mater Salutis Hospital, Legnano
  - Fondazione IRCCS - Policlinico San Matteo, Pavia
  - AUSL Della Romagna - Ospedale Santa Maria delle Croci, Ravenna
  - Istituto Clinico Humanitas, Rozzano
  - Azienda Ospedaliero - Universitaria "Santa Maria della Misericordia" di Udine, Udine
- Academisch Ziekenhuis Maastricht, Maastricht, Netherlands
- Spain (4):
  - Hospital De La Santa Creu I Sant Pau, Barcelona
  - UOMi Cancer Center, Barcelona
  - Hospital Quironsalud Sagrado Corazon, Seville
  - University Hospital Virgen del Rocio, Seville

IPD SHARING:
Plan to Share IPD: No